CLINICAL TRIAL: NCT05229276
Title: Efficacy of Sternum GuardTM in Comparison of Bone Wax in Post Cardiac Surgery Patient: A Single Blind, Single Centre, Randomized Control Trial
Brief Title: Efficacy of Sternum Guard in Post Cardiac Surgery Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Vygon GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Dudy Arman Hanafy, Sp. BTKV (K), MARS, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/402/KEP.097/2019; 1706100560 (Other: University of Indonesia - Harapan Kita National Heart Center)
Record Dates: First submitted 2021-11-09; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease; Congenital Heart Disease in Adolescence; Post Operative Wound Infection; Surgical Site Infection; Postoperative Hemorrhage
Keywords: Sternum Guard; Bone Wax; Median sternotomy; surgical site infection; operative blood loss
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Surgical Wound Infection; Postoperative Hemorrhage | interventions — bone wax

STUDY DESIGN:
Intervention Model Description: A single-blind, single center, parallel phase 4 randomized clinical trial was conducted with two intervention arms: an intervention arm with the use of Sternum GuardTM and a control arm with the use of bone wax in which the subjects' recruitment and treatment were conducted simultaneously by means of a block randomization.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects/participants were not aware of the arms/treatment given as they were under general anesthesia during the application of interventions being studied. Besides, during the informed consent for the elective sternotomy procedure, subjects were extensively given explanation of the purpose, methods, benefits and risks of the procedure including the randomized nature of the allocation to either arms of the study.
  Principal investigators as well as outcomes assessor were kept unaware of the randomization of interventions as they both were restricted for assessing the patients' medical record and the patient identity were coded in the primary database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sternum Guard (Experimental): The treatment of interest was Sternum GuardTM application during sternotomy.
  Interventions: Other: Sternum Guard
- Bone wax (Active Comparator): The 'bone wax' arm was the control group of active comparator as the widely-used materials during sternotomy.
  Interventions: Other: Bone Wax

INTERVENTIONS:
Other: Sternum Guard — The intervention being assessed is a surgical drape used as a cover of sternal bones and the neighboring structures exposed during median sternotomy named Sternum Guard.
  Sternum guard® is a single use, sterile surgical drape with modified cellulose designed specifically to reduce the risk of surgical site infection (SSI).
  It is made of 4 parts, the main part is in contact with the retractors and the sternum edge. It is made of carboxymethylated cellulose (CMC) spunlace which makes direct contact with the sternum edges. It contributes to blood absorption, to decreasing of pH environment, and to haemostatic action through a physical effect (compression); another part was made from hydrophilic spunbond (swabs) allowing blood absorption, comfort and protection
  Other Names: Sternum GuardTM, Vygon, Netherlands, product code 40.90.11
  Arms: Sternum Guard
Other: Bone Wax — patients in this group were given Bone Wax as the hemostatic material during sternotomy. Midline sternotomy with an oscillating saw was conducted after standard aseptic surgical techniques. Bone wax was applied to both spongiosa surfaces of resected sternal bones until bleeding had ceased.
  Other Names: Bone Wax, Braun Aesculap AG & CO. KG, Duisburg, Germany
  Arms: Bone wax

SUMMARY:
This is a single-center, single-blind, randomized parallel superiority trial comparing two groups; Sternum GuardTM as the treatment arm and Bone Wax as the active control group. Both investigated modalities are materials used during sternotomy for covering the sewn sternal edge. The primary outcomes of this study comprised of four parameters; namely surgical site infection (superficial or deep infection), sternal dehiscence, hemostatic effect, and surgeon's satisfaction rate. The first three primary outcomes were assessed during the operation, at the end of the hospital stay, 14 days, and 30-days postoperative.

DETAILED DESCRIPTION:
A single center randomized controlled clinical trial was conducted at Harapan Kita National Cardiovascular Center, Jakarta, Indonesia as the tertiary cardiovascular referral hospital. The RCT was conducted from May 17th, 2020 until October 20th, 2021 (current status: completed). This study assessed the efficacy of Sternum GuardTM, a commercially-available nonwoven cellulose based, single use, sterile surgical drape used for covering the dissected sternal bone edge during median sternotomy for cardiac surgery. The active comparator/ control group in this study is the use of Bone wax, a vaseline and beeswax-made materials widely used during sternotomy as a mean of bleeding control. The subjects were adults undergoing elective cardiac surgery with median sternotomy approach for any indication. Both the patients and the principal investigators were blinded for the treatment-control allocation, but the surgeon were not blinded for the materials used. The patients were purposively selected and were randomly assigned to one of the arms with block randomization. The primary outcomes of this study comprised of four parameters; namely surgical site infection (superficial or deep infection), sternal dehiscence, hemostatic effect, and surgeon's satisfaction rate. The first three primary outcomes were assessed during the operation, at the end of the hospital stay, 14 days, and 30-days postoperative. The minimum sample size was 414 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages > 18 years old
* Patients who are scheduled electively for cardiac surgery
* Cardiac surgery with the usage of cardiopulmonary bypass machine
* Patients who are agreed to participate in this study

Exclusion Criteria:

* Patients who are scheduled for surgery in emergency or urgent manner
* Patients with the history of uncontrolled hypertension and uncontrolled diabetes mellitus.
* Patients with the history of past cardiac surgery

Drop - out Criteria:

* Patients who are pronounced death on operation table
* Patients who are pronounced death within hospitalization
* Patients who are lost to follow up (Day 30 post-operative)
* Patients who are not committed for the whole stage of the research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | within 30 days after the sternotomy surgery performed
  A surgical site infection is an infection occurring within 30 days after the operation and only involving the skin and subcutaneous tissue (superficial) or involving deep soft tissues (fibrous connective tissues and muscle layers) of the post-surgical incision wounds.
  Superficial surgical site infections is identified by at least one of the following: purulent drainage, organisms isolated from an aseptically-obtained culture of fluid or tissue from the surgical site, presence of signs or symptoms of infection: pain or tenderness, localised swelling, redness or heat, or diagnosis of SSI by the surgeon or attending physician.
  A deep incisional SSI is an infection appears to be related to the operative procedure and involves deep soft tissues which is indicated by either; purulent drainage, a deep incision spontaneously dehisces, an abscess, diagnosis of a deep incisional SSI by a surgeon or attending physician.
Haemostatic effect | immediately after the median sternotomy surgery finished
  It will assess the quantity of blood lost from the sternal edges in Sternum GuardTM and Bone Wax group. The Sternum GuardTM and sterile drapes will be weighed before and after surgery to estimate the blood lost.
Satisfaction rate | within 24 hours after surgery
  A rating value from the surgeon as the user of the materials being investigated in terms of satisfaction upon the performance and practicality of the either materials from surgeon's personal opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Komite Etik of National Cardiovascular Center Harapan Kita, Study Chair — Ethical Committee of National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
the study protocol, ethical clearance letter, the primary database of the study, as well as the study's analysis plan and the manuscript of the study will be made available on the permission by the grant provider and ethical committee
Supporting Information: Study Protocol, ICF, CSR
Time Frame: November 30, 2021 for 2 (two) years
Access Criteria: for peer-reviewing or for further analysis or when needed by authors of a systematic review/meta analysis of randomized controlled trials

REFERENCES:
- [Result] Ohta S, Nishiyama T, Sakoda M, Machioka K, Fuke M, Ichimura S, Inagaki F, Shimizu A, Hasegawa K, Kokudo N, Kaneko M, Yatomi Y, Ito T. Development of carboxymethyl cellulose nonwoven sheet as a novel hemostatic agent. J Biosci Bioeng. 2015 Jun;119(6):718-23. doi: 10.1016/j.jbiosc.2014.10.026. Epub 2014 Dec 3. PMID 25488042
- [Result] Lewis KM, Spazierer D, Urban MD, Lin L, Redl H, Goppelt A. Comparison of regenerated and non-regenerated oxidized cellulose hemostatic agents. Eur Surg. 2013;45(4):213-220. doi: 10.1007/s10353-013-0222-z. Epub 2013 Jul 4. PMID 23950762
- [Result] Schonauer C, Tessitore E, Barbagallo G, Albanese V, Moraci A. The use of local agents: bone wax, gelatin, collagen, oxidized cellulose. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S89-96. doi: 10.1007/s00586-004-0727-z. Epub 2004 Jun 22. PMID 15221572
- [Result] Liu Z, Dumville JC, Norman G, Westby MJ, Blazeby J, McFarlane E, Welton NJ, O'Connor L, Cawthorne J, George RP, Crosbie EJ, Rithalia AD, Cheng HY. Intraoperative interventions for preventing surgical site infection: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2018 Feb 6;2(2):CD012653. doi: 10.1002/14651858.CD012653.pub2. PMID 29406579

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05229276/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT05229276/ICF_001.pdf